CLINICAL TRIAL: NCT05915637
Title: Investigation of Preoperative Frailty in Elderly Patients With Colorectal Cancer and Correlation Between Preoperative Frailty and Early Postoperative Prognosis
Status: Completed | Type: Observational
Sponsor: Zunyi Medical College (Other)
Responsible Party: Principal Investigator, Yongmei Zhang, Study Director, Zunyi Medical College
Other Study IDs: KLLY-2021-025
Record Dates: First submitted 2023-06-01; First posted 2023-06-23 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To investigate and analyze the status of preoperative frailty and its influencing factors in elderly patients with colorectal cancer using FRALL scale and other related scales, and to explore the correlation between preoperative frailty and early prognosis in elderly patients with colorectal cancer, so as to attract the attention of medical staff to preoperative frailty in this population and provide a preliminary research basis for the study of frailty intervention in these patients.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥60 years old;
2. Colorectal cancer was diagnosed according to the Chinese Guidelines for Diagnosis and Treatment of Colorectal Cancer (2020 edition) and planned to undergo elective laparoscopic radical resection of colorectal cancer;
3. able to complete physical assessment without communication barriers;
4. voluntarily participated in this study after informed consent.

Exclusion Criteria:

1. taking antidepressants, levodopa, donepezil hydrochloride and other drugs;
2. patients with preoperative colorectal cancer surgery or neoadjuvant therapy;
3. patients with TNM stage Ⅳ;
4. complicated with other malignant tumors except primary skin cancer or melanoma.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Colorectal cancer was diagnosed according to the Chinese Guidelines for Diagnosis and Treatment of Colorectal Cancer (2020 edition) and planned to undergo elective laparoscopic radical resection of colorectal cancer
Sampling Method: Non-Probability Sample
Enrollment: 336 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Fatigue Assessment | 7 days
  Status of frailty will be assessed by FRALL Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Yongmei Zhang, Zunyi, Guizhou, China